CLINICAL TRIAL: NCT01463501
Title: Prospective Randomized Phase Ⅱ Trial Comparing Preoperative Chemoradiotherapy (Paclitaxel and Carboplatin) Followed by Surgery to Surgery Followed by Postoperative Chemoradiotherapy (Paclitaxel and Carboplatin) for Esophageal Cancer
Brief Title: Neoadjuvant Versus Adjuvant Therapy in Treating Resectable Thoracic Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZhejiangCH09
Record Dates: First submitted 2011-08-30; First posted 2011-11-02 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2011-09

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Resectable; Neoadjuvant chemoradiotherapy; Adjuvant chemoradiotherapy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Neoadjuvant Therapy; Chemoradiotherapy, Adjuvant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant Treatment (Experimental): Preoperative chemotherapy/radiotherapy
  Interventions: Other: Neoadjuvant chemoradiotherapy
- Adjuvant Treatment (Experimental): Postoperative chemotherapy/radiotherapy
  Interventions: Other: Adjuvant chemoradiotherapy

INTERVENTIONS:
Other: Neoadjuvant chemoradiotherapy — Paclitaxel/carboplatin and concurrent radiation (50.4Gy/28f) followed by surgery, consolidate paclitaxel/carboplatin 2 cycles.
  Other Names: Neoadjuvant Treatment
  Arms: Neoadjuvant Treatment
Other: Adjuvant chemoradiotherapy — Surgery followed by paclitaxel/carboplatin and concurrent radiation (50.4Gy/28f), consolidate paclitaxel/carboplatin 2 cycles.
  Other Names: Adjuvant Treatment
  Arms: Adjuvant Treatment

SUMMARY:
This is a prospective Randomized Phase Ⅱ Trial Comparing Preoperative Chemoradiotherapy (Paclitaxel and carboplatin) Followed by Surgery to Surgery Followed by Postoperative Chemoradiotherapy (Paclitaxel and carboplatin) for Esophageal Cancer.

DETAILED DESCRIPTION:
Patient Population:

Thoracic esophageal cancer able to tolerate tri-modality therapy; Clinical stage T3-4, N0-1, M0

Scheme:

Patients are randomized to 2 arms:

Arm A:

Paclitaxel/carboplatin and concurrent radiation (50.4Gy/28f) followed by surgery, consolidate paclitaxel/carboplatin 2 cycles.

Arm B:

Surgery followed by paclitaxel/carboplatin and concurrent radiation (50.4Gy/28f), consolidate paclitaxel/carboplatin 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell carcinoma or adenocarcinoma of the thoracic esophagus (> 20cm from the incisors) or gastroesophageal junction are included.
* No distant metastases (M0).
* Patients will be stratified by stage (clinical N0 versus clinical N1).
* Patients with tumours within 3 cm distal spread into gastric cardia as detected by esophagogastroscopy.
* Resectable mediastinal nodes are eligible.
* No prior chemotherapy for this malignancy.
* No prior radiotherapy that would overlap the field(s) treated in this study.
* Patients with other malignancies are eligible only if > 5 years without evidence of disease or completely resected or treated non-melanoma skin cancer.
* Age > 18 years and able to tolerate tri-modality therapy at the discretion of the treating thoracic surgeon, medical and radiation oncologists. Tumours must be resectable after assessment by the thoracic surgeon.

Exclusion Criteria:

* Cancers of the cervical esophagus (< 20 cm are excluded).
* Tumours that have > 3 cm of spread into cardia of the stomach are considered gastric cancers and are ineligible.
* Patients with biopsy (by endoscopic ultrasound, laparoscopy, or laparotomy ) proven metastatic supraclavicular nodes are ineligible.
* Patients with biopsy proven metastatic celiac nodes are ineligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Scores of Quality of life | 1 year
  Assess the quality of life based on FACT-E.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 year
  Assess the safety and tolerability based on NCI CTC V4.0

SECONDARY OUTCOMES:
Disease-free Survival | 3 years
  Three years disease free survival will be evaluated.
Overall Survival | 3 years
  Three years overall survival will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Weimin Mao, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China